CLINICAL TRIAL: NCT03658525
Title: Prostate Radiotherapy Integrated With Simultaneous MRI (The PRISM Study)
Acronym: PRISM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCR4888
Record Dates: First submitted 2018-08-06; First posted 2018-09-05 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-08

CONDITIONS: Prostate Cancer
Keywords: MR GUIDED RADIOTHERAPY
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: To assess delivery of prostate IMRT on the MR linac
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MR LINAC RADIOTHERAPY (Experimental): RADIOTHERAPY DELIVERED ON MR LINAC
  Interventions: Device: MR LINAC

INTERVENTIONS:
Device: MR LINAC — MR GUIDED PROSATE RADIOTHERAPY

SUMMARY:
Currently radiotherapy for prostate cancer is directed using scans or X-Rays, which ensures the radiotherapy treatment 'hits the target' and avoids the healthy tissues around the prostate. There are two current methods of radiotherapy image guidance- either placing small gold seeds into the prostate and taking XRays or doing a small CT scan of the prostate region each day. Neither of these methods are perfect and have drawbacks and inaccuracies.

The best way to see the prostate is with an MRI scan - this shows the edge of the prostate much more clearly and can even show the area of most aggressive cancer within the prostate. Shortly the investigators will have the ability to use a new machine - an MR-Linac - which combines an MR scanner and a radiotherapy machine.

As well as giving the investigators a clearer picture, and enabling the investigators to keep watching the prostate while the participant has their treatment (not currently possible with standard machines) this new machine will also allow the investigators to change the radiotherapy plan if they can see that the internal anatomy has shifted day to day. Currently the investigators have to give the same radiotherapy plan each day, which means the investigators have to treat a 'safety margin' around to prostate to allow for these day to day anatomy changes (e.g. rectal filling).

The aim of this study is to assess the technical feasibility of delivering radical radiotherapy for prostate cancer using the MR-Linac, including the feasibility of changing the radiotherapy plan on a daily basis to mirror internal anatomy changes. The investigators will recruit 30 patients with localised prostate cancer who need radiotherapy. The team will deliver the same dose in the same number of days i.e. the same as standard radiotherapy. Side effects will also be assessed by physicians and using patient questionnaires.

ELIGIBILITY:
Inclusion Criteria:

All of the following criteria should be met for study entry.

* Histologically confirmed adenocarcinoma prostate- grade group 3 or less (Gleason 4+3=7 or less).
* Staging T2-T3a,N0M0 (MRI or DRE staging allowed).
* PSA<25.
* 6 months short course androgen deprivation therapy allowed, not mandated.
* Maximum prostate volume 70cc.
* IPSS <12 at baseline.
* WHO performance status 0 or 1.
* Written informed consent.

Exclusion Criteria:

If one of the following criteria are met, the patient is not eligible for the study

* Other invasive malignancy within the last two years- excluding basal cell carcinoma and squamous cell carcinoma of the skin.
* Patients who, in the opinion of the Local PI, require long course (> 6 months) ADT.
* Contraindications to MRI.Including pacemaker, implanted devices, any non-MR compatible metallic implants.Severe claustrophobia.
* Contraindications to gold fiducial marker implantation.Clotting disorders, very high risk of bleeding.Clinically unacceptable risk of temporarily stopping anticoagulation or antiplatelet medications.
* Contraindications to prostate radiotherapy,Previous pelvic radiotherapy.Clinically significant inflammatory bowel disease.
* Bilateral or single hip replacements.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — INVOLVES PROSTATE CANCER PATIENTS SO MUST BE MALE
Enrollment: 30 (Estimated)
Dates: Start 2018-08-07 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients in whom the imaging and treatment on the MR Linac (i.e. total time on the treatment couch) can be completed within 1 hour on 90% of fractions as assessed by the radiotherapy timing sheet. | 2 YEARS
  The radiotherapy timing sheet will be used to record the length of time for patients to have their MR guided adaptive radiotherapy for each fraction. This information will then inform if treatment can be given in a clinically feasible time frame.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Marsden - Surrey, Sutton, England, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
ANONYMISED DATA WILL BE SHARED WITHIN THE ELEKTA CONSORTIUM